CLINICAL TRIAL: NCT02953951
Title: Blood Transfusions May Impair Endothelium-dependent Vasodilatation in Isolated Left Mammary Arterial Artery Rings and Peripheral Artery Tonometry During Coronary Artery Bypass Surgery
Brief Title: Blood Transfusions in Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alessio Rungatscher, MD, PhD, FAHA, Universita di Verona
Other Study IDs: CIRSAL-1231
Record Dates: First submitted 2016-10-16; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-10

CONDITIONS: Excessive Amount of Blood / Fluid Transfusion
Keywords: blood transfusion; free hemoglobin; nitric oxide; endothelium-dependent vasodilatation; peripheral artery tonometry; cardiac surgery.
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, left internal mammary artery (discared rings)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stored Blood Cells: Blood transfusion:
  Stored blood cells transfused patients
  Interventions: Other: blood transfusion
- Autologous Salvaged Blood: Blood transfusion:
  Autologous salvaged blood transfused patients
  Interventions: Other: blood transfusion
- Control: Blood transfusion:
  No transfusion patients

INTERVENTIONS:
Other: blood transfusion — blood transfusion different sources
  Groups: Autologous Salvaged Blood; Stored Blood Cells

SUMMARY:
The hemolytic product free-hemoglobin (fHb) reduces nitric oxide (NO) bioavailability. The present study aims to establish whether transfusions of stored allogenic blood or intraoperative autologous salvaged blood result in increased circulating fHb levels and NO consumption with effects on arterial NO-dependent blood flow measured in isolated left mammary artery rings and by peripheral artery tonometry in patients undergoing CABG surgery.

DETAILED DESCRIPTION:
Introduction

Several studies have implicated red blood cell (RBC) transfusion as a risk factor for increased morbidity as well as short- and long-term mortality after coronary artery bypass graft surgery (CABG). Interestingly, this effect is most pronounced among patients undergoing isolated CABG, suggesting that a harmful mechanism of RBC transfusion is not generalizable to all types of surgical procedures but instead may be specific to those patients.

The mechanisms by which blood transfusion may contribute to organ injury, dysfunction and death remain uncertain. Besides the quantity of RBC transfusions, the quality of the product has also been associated with differences in mortality and morbidity.

The use of intraoperative cell salvage and autologous blood transfusion has become an important method of blood conservation. The main aim of autologous transfusion is to reduce the need for allogeneic blood transfusion and its associated complications. However hemolysis and high cell-free hemoglobin (fHb) contents are associated with cell washing devices that collect anticoagulated shed or recovered blood, wash and separate the RBC by centrifugation, and re-infuse the RBC.

fHb is a potent scavenger of nitric oxide (NO), which mediates endothelium-dependent vasodilation, and may therefore be responsible for microvascular perfusion disturbances (arterial spasm). Indeed endothelial dysfunction and persistent microvascular alterations are associated with organ failure and death.

Increasing hemolysis and release of fHb were also documented as a function of time during prolonged RBC storage. Transfusion of RBC stored for less than 14 days has been associated with favourable outcomes when compared with transfusion of RBC stored for a prolonged time. Changes in red cell structure and function during blood banking and storage have been referred to as the red cell storage lesion.

The present study aimed to assess whether transfusion of stored allogeneic blood or intraoperative autologous salvaged blood results in differently increased circulating fHb levels and plasma NO consumption with effects on arterial NO-dependent blood flow in patients undergoing CABG surgery.

Methods

Study design This single-centre, prospective observational cohort study was based on consecutive patients undergoing elective isolated CABG with cardiopulmonary bypass (CPB) at our institution between January 2014 and May 2014. Perioperative and postoperative data were collected prospectively. The study protocol was approved by the Institution's Ethical Committee/Institutional Review Board.

Surgery Anaesthesia was standardized and maintained with propofol, sufentanil and vecuronium. Surgery was always performed through median sternotomy. LIMA was harvested as a pedicle, anastomosed to the left anterior descending artery in all cases, and never used as a free graft. CPB circuit included a Sorin phosphorylcholine-coated tubing set (Sorin Group SpA, Milano, Italy), a Jostra roller pump (Jostra, Maquet Cardiopulmonary, Hirrlingen, Germany), and a hollow fiber membrane coated oxygenator, which incorporated also a 40 μm filter (Sorin Synthesis™, Sorin Group Spa, Milano, Italy). Heparin was given at a dose of 300 IU/kg to achieve a target activated clotting time of 480 s or above. The extracorporeal circuit was primed with 1400 mL of Ringer's lactate solution and 5000 IU of heparin. A non-pulsatile CPB flow was established at 2.4 L/min. Buckberg crystalloid cardioplegic solution was used to maintain cardioplegia during aortic cross-clamping. Infusion of 4 mg/kg of protamine was used to neutralize heparin after finishing the CPB. Residual blood was sucked from the venous reservoir into the cell saver collection reservoir using a dual lumen tube connected to a vacuum pump and subsequently transferred to the 125-ml centrifuge bowl of the cell saver (Cell Saver 5; Haemonetics, Braintree, MA, USA). Cells were washed using 2000 ml bags NaCl 0.9% with 30.000 IU of heparin (Athena Pharma, Rome, Italy). The following cell saver program was used for the cell saver: 5600 r.p.m., filling and washing rate of 250 ml/min, emptying rate 250 ml/min, wash volume 1000 ml. Concentrated blood cells were drained into a patient labelled soft collection bag.

Transfusion protocol Transfusion of packed RBC was indicated at Hb levels < 7 g/l during CPB. After the end of CPB an Hb level < 9 g/l indicated requirement of autologous salvaged concentrated blood cells and/or packed RBC.

ELIGIBILITY:
Inclusion Criteria:

* elective CABG surgery

Exclusion Criteria:

* vasopressors/inotropes during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing elective isolated CABG with cardiopulmonary bypass (CPB) at our institution between January 2014 and May 2014.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in free hemoglobin plasma level (mg/dl) | 1) beginning of surgery, 2) after 12 hours
  analyzed by derivative spectrometry

SECONDARY OUTCOMES:
Endothelium-dependent arterial relaxation (in vitro) | after 12 hours
  arterial rings assay
Endothelium-dependent arterial relaxation (in vivo) | after 12 hours
  Peripheral artery tonometry
Change in Nitric oxyde consumption (umol/l) | 1) beginning of surgery, 2) after 12 hours
  Nitric Oxide Analyzer (Sievers)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Rungatscher, MD, PhD, Principal Investigator — Universita di Verona
Locations (1):
- Azienda Ospedalieva Universitaria Integrata, Verona, Italy

IPD SHARING:
Plan to Share IPD: No